CLINICAL TRIAL: NCT05550038
Title: Diagnostic Performance of General Practitioners in Compression Ultrasound for the Diagnosis of Proximal Deep Vein Thrombosis of the Lower Limbs
Brief Title: Diagnostic Performance of General Practitioners in Compression UltraSound
Acronym: GPCUS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of inclusions
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-0114; 22.02437.000091 (Other: CPP OUEST II); 2022-A01244-39 (Other: ANSM)
Record Dates: First submitted 2022-09-08; First posted 2022-09-22 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-01

CONDITIONS: Deep Vein Thrombosis
Keywords: DVT; Vein thrombosis; Thrombophlebitis
MeSH Terms: conditions — Venous Thrombosis; Thrombophlebitis

STUDY DESIGN:
Intervention Model Description: All included patients will have a compression ultrasound performed by the general practitioner followed within 72 hours by a whole leg ultrasound with Doppler performed by the vascular physician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- compression ultrasound (Experimental): All patients receive a 3-point compression ultrasound followed within 72 hours by a whole-leg ultrasound with Doppler performed by a vascular physician.
  Interventions: Diagnostic Test: Compression ultrasound

INTERVENTIONS:
Diagnostic Test: Compression ultrasound — Patients receive a 3-point compression ultrasound performed by the general practitioner to look for proximal deep vein thrombosis.
  Other Names: three-point compression; three-point compression ultrasound; three-point point-of-care ultrasound technique

SUMMARY:
The objective of this study is to evaluate the diagnostic efficiency of general practitioners for the diagnosis of proximal deep vein thrombosis of the lower limbs compared with whole-leg ultrasound with Doppler performed by the vascular physician.

DETAILED DESCRIPTION:
After being informed about the study and the potential risks, all patients who have given their written consent and who meet the eligibility criteria will benefit from a 3-point compression ultrasound performed by the general practitioner before being referred for a whole-leg ultrasound with Doppler at the vascular physician.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Management by a general practitioner trained in 3-point venous ultrasound
* Suspicion of deep vein thrombosis by the general practitioner with prescription of a whole-leg Doppler ultrasound by a vascular physician. It is noted that the patient can be included from the moment the general practitioner had planned to refer the patient to the vascular physician for a suspicion of DVT, including in the absence of realization of DDimer on a low probability of DVT. It may also be included in case of positive DDimer tests.
* Signed written consent
* Patient covered by the French social security system

Exclusion Criteria:

* Whole leg ultrasound performed more than 72 hours after the initial examination
* History of homolateral deep vein thrombosis
* Patient objecting to the use of his data
* Refusal of written and signed consent

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of 3 point venous compression | 72 hours
  The diagnostic performance (Sensitivity, Specificity, Positive Predictive Value, Negative Predictive Value) of 3-point venous compression ultrasound performed by general practitioners for the diagnosis of proximal venous thrombosis of the lower limbs compared to the usual recommended examination (whole leg ultrasound by a vascular physician)

SECONDARY OUTCOMES:
The evaluation of the feasibility of venous compression ultrasound in the office by the general practitioner. | 72 hours
  For each patient, the general practitioner must say whether or not he or she was successful in performing the compression ultrasound.
  The measure will be the percentage of ultrasound examinations considered successful by general practitioners.
Duration of the ultrasound performed by the general practitioner in minutes. | 72 hours
  Duration of the ultrasound performed by the general practitioner in minutes.
The interpretability of ultrasound images by general practitioners | 72 hours
  The interpretability of ultrasound images by general practitioners. For each patient, the general practitioner must note the result of his or her ultrasound (compressibility or total incompressibility of the veins on the 3 points studied). He must also correctly interpret the ultrasound result (presence of venous thrombosis in case of total incompressibility of the vein or absence of thrombosis in case of total compressibility of the vein).
  The measure will be the percentage of correct interpretation of the compression test.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas DELOMAS, Dr, Principal Investigator — Hospital Saint Lo
Locations (19):
- France (19):
  - Bayeux, Bayeux, Normandy
  - Avranches, Avranches
  - Bain de Bretagne, Bain-de-Bretagne
  - Colombelles, Colombelles
  - Condé sur vire, Condé-sur-Vire
  - Honfleur, Honfleur
  - Ifs, Ifs
  - Le Chesnay, Le Chesnay
  - Le pont de montvert, Le Pont-de-Montvert
  - Lons-le-Saunier, Lons-le-Saunier
  - Le Molay Littry, Molay
  - Ouistreham, Ouistreham
  - Paris rue de Rome, Paris
  - Percy, Percy
  - Ploerdut, Ploërdut
  - Potigny, Potigny
  - Saix, Saïx
  - Sannerville, Sannerville
  - Troarn, Troarn

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mumoli N, Vitale J, Giorgi-Pierfranceschi M, Sabatini S, Tulino R, Cei M, Bucherini E, Bova C, Mastroiacovo D, Camaiti A, Palmiero G, Puccetti L, Dentali F; PRACTICUS Study Investigators. General Practitioner-Performed Compression Ultrasonography for Diagnosis of Deep Vein Thrombosis of the Leg: A Multicenter, Prospective Cohort Study. Ann Fam Med. 2017 Nov;15(6):535-539. doi: 10.1370/afm.2109. PMID 29133492
- [Background] Mumoli N, Vitale J, Cocciolo M, Cei M, Brondi B, Basile V, Sabatini S, Gambaccini L, Carrara I, Camaiti A, Giuntoli S, Dentali F. Accuracy of nurse-performed compression ultrasonography in the diagnosis of proximal symptomatic deep vein thrombosis: a prospective cohort study. J Thromb Haemost. 2014 Apr;12(4):430-5. doi: 10.1111/jth.12522. PMID 24495051
- [Background] Pomero F, Dentali F, Borretta V, Bonzini M, Melchio R, Douketis JD, Fenoglio LM. Accuracy of emergency physician-performed ultrasonography in the diagnosis of deep-vein thrombosis: a systematic review and meta-analysis. Thromb Haemost. 2013 Jan;109(1):137-45. doi: 10.1160/TH12-07-0473. Epub 2012 Nov 8. PMID 23138420
- [Background] Lee JH, Lee SH, Yun SJ. Comparison of 2-point and 3-point point-of-care ultrasound techniques for deep vein thrombosis at the emergency department: A meta-analysis. Medicine (Baltimore). 2019 May;98(22):e15791. doi: 10.1097/MD.0000000000015791. PMID 31145304